CLINICAL TRIAL: NCT06036238
Title: Innovative Strategies to Promote Biomedical HIV Prevention Uptake and Retention Among High-risk Adults at Drinking Venues in Kenya and Uganda
Brief Title: The Outreach and Prevention at ALcohol Venues in East Africa Study (OPAL-East Africa- Aim 2) (OPAL-Aim 2)
Acronym: OPAL-Aim 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Berkeley (Other); Makerere University (Other); Infectious Diseases Research Collaboration, Uganda (Other); Kenya Medical Research Institute (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-37054-2; 1R01AA030464-01 (NIH)
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: HIV/AIDS
Keywords: Alcohol use; Biomedical HIV prevention; Uganda; Kenya; Counseling intervention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Alcohol Drinking | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Control) (Active Comparator): Standard of care; alcohol counseling per Ministry of Health (MoH) guidelines
  Interventions: Behavioral: Standard of Care
- Healthy Living Intervention (Experimental): Healthy Living Intervention in-person alcohol counseling with booster phone calls
  Interventions: Behavioral: Healthy Living Intervention (HLI)

INTERVENTIONS:
Behavioral: Healthy Living Intervention (HLI) — The Healthy Living Intervention (HLI) is a brief alcohol counseling intervention developed using the Information, Motivation, and Behavioral skills (IMB) model, a framework in which information, motivation, and behavioral skills are key determinants of health behavior. Participants initiating PrEP will be randomized to either HLI or standard of care alcohol counseling.
  Arms: Healthy Living Intervention
Behavioral: Standard of Care — Participants who are randomized to the control arm will receive basic alcohol counseling through the Ministry of Health if it is provided as standard of care.
  Arms: Standard of Care (Control)

SUMMARY:
This study will evaluate the effect of a brief alcohol counseling intervention on PrEP and PEP adherence among adults with heavy alcohol use at high risk for HIV, while gaining insights into the facilitators, barriers, and cost-effectiveness of this approach.

DETAILED DESCRIPTION:
The investigators have developed a mobilization strategy of integrating HIV testing within multi-disease screening to recruit >2,000 people from drinking venues in Kenya and Uganda and invite them to begin biomedical HIV prevention if eligible (OPAL Aim 1; NCT05862857)

Following uptake of biomedical HIV prevention, persons with heavy alcohol use face challenges with retention in care and adherence to PrEP/PEP. The investigators have adapted a brief alcohol counseling intervention (Health Living Intervention) to reduce alcohol use and promote antiretroviral therapy (ART) adherence and HIV viral suppression among persons with HIV in Kenya and Uganda. The investigators now need to determine whether this intervention can promote retention in biomedical prevention and PrEP/PEP adherence among adults with heavy alcohol use.

Specific Aims:

* Determine the efficacy of the Healthy Living Intervention (HLI) to reduce heavy alcohol use vs. standard care (control) on retention in biomedical HIV prevention in a randomized trial among adults with heavy alcohol use.
* Determine the cost-effectiveness of interventions that increase biomedical HIV prevention retention among adults at high-risk for HIV who attend drinking venues.

The proposed research will address the critical intersection of alcohol use and HIV risk in SSA, by promoting retention of biomedical HIV prevention and exploring associated facilitators and barriers.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years)
* HIV-uninfected (by rapid HIV antibody test)
* AUDIT-C score of >=4 for men and >=3 for women
* Attending a clinical visit for initiation of biomedical HIV prevention with oral or injectable PrEP or oral PEP (or the dapivirine vaginal ring, if available)
* Has access to a mobile phone

Exclusion Criteria:

* Ineligible for PrEP based on MoH guidelines
* Intention to move away from the study community in the coming year
* Gross inebriation or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of follow up time on biomedical prevention with PrEP or PEP | Measured 24 weeks after PrEP or PEP initiation
  The proportion of time during the 24 weeks after PrEP/PEP initiation that a person is protected from HIV with PrEP/PEP, assessed by prescription refill data. Prescription refill data will be collected from MoH medical and pharmacy records, augmented by OPAL case report forms.

SECONDARY OUTCOMES:
Proportion of follow up time on biomedical prevention with PrEP or PEP- 48 weeks | Measured over 48 weeks after PrEP or PEP initiation
  Secondary analysis of the primary outcome will measure the proportion of time that a person is protected from HIV with PrEP/PEP over 48 weeks, with integrated drug levels measured in hair samples collected at 48 weeks.
Proportion of participants with unhealthy alcohol use (defined by AUDIT-C ≥3 for women, ≥4 for men, and phosphatidylethanol (PEth) ≥50 ng/mL) at week 48 | Measured 48 weeks after PrEP or PEP initiation
  Study staff will assess AUDIT-C scores (modified to refer to the prior 3 months, with a minimum of 0, indicating no alcohol use, and a maximum of 12) with a standard drink guide adapted to local context at baseline and every 12-weeks post-baseline. Blood will also be collected, and dried blood spots prepared for phosphatidylethanol (PEth) testing (measured in ng/mL with higher levels associated with greater alcohol use) at baseline and 48-weeks for confirmation of self-reported alcohol use.
Proportion of participants with HIV seroconversion by week 48 | Measured 48 weeks after PrEP or PEP initiation
  HIV seroconversion will be measured as documented rapid HIV antibody test positivity with Geenius confirmation or documented detectable HIV viral load, with rapid HIV testing. HIV testing will occur at PrEP refill and injection visits, or completion of a course of PEP.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Chamie, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (2):
- Kenya Medical Research Institute (KEMRI), Mbita, Kenya
- Infectious Diseases Research Collaboration (IDRC), Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Per the approved Data Sharing agreement with the NIAAA Data Archive, the investigators will share de-identified IPD from our baseline questionnaire, which includes questions about subject demographics, HIV risk, and alcohol use.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 3 months after article publication and the data will be made accessible for up to 36 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP).